CLINICAL TRIAL: NCT06127628
Title: Effectiveness of Ultrasound-guided Scalp Block for Supratentorial Craniotomy: a Randomised Controlled Trial
Brief Title: Effectiveness of Ultrasound-guided Scalp Block for Supratentorial Craniotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Malaysia Sarawak (Other)
Responsible Party: Principal Investigator, Samuel Ern Hung Tsan, Clinical lecturer, University Malaysia Sarawak
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRR ID-23-03179-N5K
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Pain, Postoperative; Anesthesia
Keywords: Scalp block; Pain; Supratentorial craniotomy; Ultrasound
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: Parallel groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of participants and outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided scalp with ropivacaine 0.375% (Experimental): Ultrasound-guided scalp block performed for supraorbital nerve, supratrochlear nerve, zygomaticotemporal nerve, auriculotemporal nerve, superficial cervical plexus, greater occipital nerve and third occipital nerve. The local anaesthetic used will be ropivacaine 0.375%.
  Interventions: Procedure: Ultrasound-guided scalp block with ropivacaine 0.375%
- Standard treatment (No Intervention): Standard perioperative anaesthetic and surgical treatment will be performed, with the omission of ultrasound-guided scalp block

INTERVENTIONS:
Procedure: Ultrasound-guided scalp block with ropivacaine 0.375% — Scalp block will be performed under USG guidance, using the technique described by Tsan et al. The block needle used will be an echogenic block needle, with a length of 50 mm, and a diameter of 22 G. Trained personnel comprising of the investigators in this study will perform the scalp block. Using ultrasound to identify landmarks, ropivacaine 0.375% will be administered in volumes of 1.5 ml to 3 ml. The nerves targeted will be the supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, greater auricular, lesser occipital, greater occipital and third occipital nerves.
  Arms: Ultrasound-guided scalp with ropivacaine 0.375%

SUMMARY:
Pain management in patients undergoing neurosurgery is a very important issue. The effectiveness of USG-guided scalp blocks for pain management in craniotomy surgery is currently not known. The purpose of this clinical trial is to evaluate the effectiveness of ultrasound-guided scalp block when performed in patients who undergo supratentorial craniotomies.

DETAILED DESCRIPTION:
The main research questions this trial will answer are:

1. In patients undergoing elective supratentorial craniotomy under general anaesthesia, does USG-guided scalp block affect postoperative pain compared to standard treatment?
2. In patients undergoing elective supratentorial craniotomy under general anaesthesia, does USG-guided scalp block affect postoperative opioid consumption compared to standard treatment?
3. In patients undergoing elective supratentorial craniotomy under general anaesthesia, does USG-guided scalp block affect intraoperative haemodynamic parameters (blood pressure and heart rate) compared to standard treatment?

This clinical trial compares ultrasound-guided scalp block with ropivacaine 0.375% versus standard treatment.

The findings of this clinical trial may potentially revolutionise the practice of regional anaesthesia and analgesia in intracranial surgeries. This will lead to better patient outcomes by improving the perioperative care of patients undergoing craniotomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* All American Society of Anesthesia class I to III patients undergoing elective supratentorial craniotomies under general anaesthesia.

Exclusion Criteria:

1. Refusal to participate in the study
2. Contraindications to the performance of scalp block, such as local infections
3. Allergy to ropivacaine hydrochloride
4. Age < 18 years old
5. Undergoing emergency craniotomies, posterior fossa surgery, or burr holes surgery
6. Pre-existing chronic pain (defined as persistent or recurrent pain lasting > 3 months)
7. History of drug addiction (illicit substances and opioids use) or chronic alcohol abuse
8. Presence of uncontrolled systemic arterial hypertension, severe cardiovascular disease, severe kidney or severe liver diseases
9. Predicted to require postoperative ventilation in the intensive care unit
10. Psychiatric disorders, serious neurological diseases, or reduced consciousness GCS < 14

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Pain scores will be measured at 1, 6, 24, and 48 hours after surgery.
  Postoperative pain as measured by the visual analogue scale, with no pain being 0 and the maximal pain possible being 10.

SECONDARY OUTCOMES:
Opioid consumption postoperatively | Measured at 24 and 48 hours after surgery
  Overall postoperative morphine-equivalent consumption
Intraoperative blood pressure stability during stimulating points of surgery | Measurements will be made at time 0 (before stimulation), time-1 (1 minute after stimulation), time-3 (3 minutes after stimulation) and time-5 (5 minutes after stimulation).
  Mean arterial pressures in mmHg at skull-pinning, skin incision and craniotomy.
Intraoperative heart rate stability during stimulating points of surgery | Measurements will be made at time 0 (before stimulation), time-1 (1 minute after stimulation), time-3 (3 minutes after stimulation) and time-5 (5 minutes after stimulation).
  Heart rates in beats per minute at skull-pinning, skin incision and craniotomy.

OTHER OUTCOMES:
Complications of ultrasound-guided scalp block | Within 48 hours after procedure
  Adverse events
Postoperative nausea and vomiting | Within 48 hours after surgery
  Incidence and severity of postoperative nausea and vomiting
Patient satisfaction with pain management | Within 48 hours after surgery
  Satisfaction of participants postoperatively regarding quality of pain management, as measured with Likert scale, 5 being maximal satisfaction, 1 being least satisfaction.
Intraoperative anaesthetic usage | During surgery
  Amount of intraoperative anaesthetic agents used
Complications associated with opioid usage | Within 48 hours after surgery
  Complications such as pruritus, respiratory depression, sedation, urinary retention, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Sarawak General Hospital, Kuching, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsan SEH, Goh CH, Tan PCS. Ultrasound-Guided Scalp Blocks for an Awake Craniotomy: A Case Report. A A Pract. 2022 Sep 20;16(9):e01618. doi: 10.1213/XAA.0000000000001618. eCollection 2022 Sep 1. PMID 36136961